CLINICAL TRIAL: NCT00354185
Title: A Phase I Study of PXD101 in Combination With 17-AAG in Advanced Malignancies
Brief Title: PXD101 and 17-N-Allylamino-17-Demethoxygeldanamycin in Treating Patients With Metastatic or Unresectable Solid Tumors or Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00006; CO 05906; WCCC-CO-05906; NCI-7277; U01CA062491 (NIH)
Record Dates: First submitted 2006-07-19; First posted 2006-07-20 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-05

CONDITIONS: Adult Nasal Type Extranodal NK/T-cell Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Intraocular Lymphoma; Nodal Marginal Zone B-cell Lymphoma; Post-transplant Lymphoproliferative Disorder; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; Stage III Adult Burkitt Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Mixed Cell Lymphoma; Stage III Adult Diffuse Small Cleaved Cell Lymphoma; Stage III Adult Hodgkin Lymphoma; Stage III Adult Immunoblastic Large Cell Lymphoma; Stage III Adult Lymphoblastic Lymphoma; Stage III Adult T-cell Leukemia/Lymphoma; Stage III Cutaneous T-cell Non-Hodgkin Lymphoma; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage III Marginal Zone Lymphoma; Stage III Mycosis Fungoides/Sezary Syndrome; Stage III Small Lymphocytic Lymphoma; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Hodgkin Lymphoma; Stage IV Adult Immunoblastic Large Cell Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Adult T-cell Leukemia/Lymphoma; Stage IV Cutaneous T-cell Non-Hodgkin Lymphoma; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Mycosis Fungoides/Sezary Syndrome; Stage IV Small Lymphocytic Lymphoma; Unspecified Adult Solid Tumor, Protocol Specific; Waldenström Macroglobulinemia
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Intraocular Lymphoma; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia | interventions — tanespimycin; belinostat

ARMS (1):
- Treatment (tanespimycin, belinostat) (Experimental): Patients receive 17-AAG IV over 2 hours on days 1, 4, 8, and 11 and PXD101 IV over 30 minutes on days 1-5. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of 17-AAG and PDX101 until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Up to 12 patients are treated at the MTD.
  Patients undergo blood collection on days 1 and 4 of course 1 for pharmacokinetic studies.
  Interventions: Drug: tanespimycin; Drug: belinostat; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: tanespimycin — Given IV
  Other Names: 17-AAG
Drug: belinostat — Given IV
  Other Names: PXD101
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I trial is studying the side effects and best dose of giving PDX101 together with 17-AAG in treating patients with metastatic or unresectable solid tumors or lymphoma. PDX101 may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the cancer. Drugs used in chemotherapy, such as 17-N-allylamino-17-demethoxygeldanamycin (17-AAG), work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving PXD101 together with 17-AAG may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability of PXD101 and 17-AAG administered to patients with refractory solid tumor malignancies.

II. To determine the maximum tolerated dose (MTD) and recommended phase II dose of PXD101 and 17-AAG in patients with refractory solid tumor malignancies.

SECONDARY OBJECTIVES:

I. To evaluate the pharmacokinetics of PXD101 and 17-AAG in patients receiving this combination.

II. To evaluate the antitumor activity of this combination, per tumor measurements using the RECIST criteria.

TERTIARY OBJECTIVES:

I. To evaluate the effect of treatment with PXD101 and 17-AAG on the transcriptional upregulation of targeted genes in tumor and surrogate tissue (PBMCs) by means of RTPCR and incorporation of the chromatin immunoprecipitation assay.

II. To evaluate the effect of this combination treatment on the post translational modification of histones from tumor and surrogate tissue (PBMCs).

OUTLINE: This is a dose-escalation study.

Patients receive 17-N-allylamino-17-demethoxygeldanamycin (17-AAG) IV over 2 hours on days 1, 4, 8, and 11 and PXD101 IV over 30 minutes on days 1-5. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of 17-AAG and PDX101 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Up to 12 patients are treated at the MTD.

Patients undergo blood collection on days 1 and 4 of course 1 for pharmacokinetic studies.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 36 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed malignancy (solid tumor or lymphoma) that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective
* Patients may have received prior treatment with either any HDAC inhibitor therapy or 17AAG, as long as they did not experience dose limiting toxicity (DLT) with these prior treatments; DLTs include

  * Toxicity: neutrophils; DLT: grade 4 toxicity (< 500/μL) for >= 7 days
  * Toxicity: febrile neutropenia; DLT: ANC < 1000/μL of any duration accompanied by fever >= 38.5ºC
  * Toxicity: platelets; DLT: grade 4 toxicity (< 25,000/μL) for >= 7 days or of any duration if accompanied by clinically significant bleeding
  * Toxicity: non-hematologic; DLT: >= grade 3 as per NCI Common Terminology Criteria for Adverse Events, Version 3.0** (except alopecia); ** for nausea and vomiting, grade 3 toxicity with maximal anti-emetic treatment will be considered dose-limiting; grade 3 diarrhea in spite of maximal anti-diarrheal therapy will be considered dose-limiting; hypersensitivity reactions to 17AAG will not be considered a DLT; asymptomatic grade 3 hypophosphatemia will not be considered a DLT
  * Toxicity: cardiac; DLT: ≥ grade 3 QTc prolongation
* ECOG performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 12 weeks
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 75,000/mcL
* Total bilirubin within normal institutional limits
* AST(SGOT)/ALT(SGPT) =< 2.5 X institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Eligibility of patients receiving any medications or substances known to affect or with the potential to affect the activity or pharmacokinetics of PXD101 or 17AAG will be determined following review of their case by the Principal Investigator or Study Chair; efforts should be made to switch patients who are taking enzyme-inducing anticonvulsant agents to other medications
* The effects of PXD101 and 17AAG on the developing human fetus are unknown; for this reason and because HDAC inhibitors as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* Within 4 weeks of first treatment: Left ventricular ejection fraction ≥ 45% per nuclear cardiac imaging or echocardiography

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered (≤ grade 1) from clinically significant adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to PXD101; there are no known allergic reactions attributed to compounds of similar chemical or biological composition to 17AAG; patients with known egg allergy should be excluded as the agent is diluted in EPL diluent
* Patients should not have taken valproic acid, another histone deacetylase inhibitor, for at least 2 weeks prior to enrollment
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because PXD101 is an HDAC inhibitor with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with PXD101, breastfeeding should be discontinued if the mother is treated with PXD101; these potential risks may also apply to other agents used in this study
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with PXD101; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* History of allergic reactions to eggs
* Patients who have significant cardiac disease including heart failure that meets New York Heart Association (NYHA) class III and IV definitions, history of myocardial infarction within 12 months of study entry, ischemic or severs valvular heart disease, uncontrolled dysrhythmias, uncontrolled hypertension, a condition requiring anti-arrhythmic therapy, or poorly controlled or unstable angina pectoris
* Patients who have a history of serious ventricular arrhythmia (VT or VF, >= 3 beats in a row) or QTc >= 450 msec for men and 470 msec for women or a history of long QT Syndrome
* Patients taking concomitant medications that prolong or may prolong QTc or may cause Tosade des Pointes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-05; Primary Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD), based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v3.0 | Up to 21 days
Number and severity of toxicity incidents, based on the NCI CTCAE v3.0 | Up to 2 years
  Dose-toxicity relationship may be explored by performing exact logistic regression analysis.

SECONDARY OUTCOMES:
Cmax (observed maximum plasma concentration) | Day 4
  Summarized by dose level with simple summary statistics. Jonckheere-Terpstra trend test will be performed. Scatterplots will be used.
Tmax (time to Cmax) | Day 4
  Summarized by dose level with simple summary statistics.
AUC0-lqc (the area under the plasma concentration-time curve as determined by the linear trapezoidal rule and where lqc is last quantifiable concentration) | Day 4
  Summarized by dose level with simple summary statistics. Jonckheere-Terpstra trend test will be performed. Scatterplots will be used.
AUC0-omega (the area under the plasma concentration-time curve from time 0 to infinity as determined by AUC0-lqc + lqc/-omega) | Day 4
  Summarized by dose level with simple summary statistics. Jonckheere-Terpstra trend test will be performed. Scatterplots will be used.
T1/2 (the terminal disposition half-life calculated as ln(2)/-beta) | Day 4
  Summarized by dose level with simple summary statistics.
CL where the clearance is calculated by dividing the total dose by AUC0-omega | Day 4
  Summarized by dose level with simple summary statistics.
Anti-tumor response (progressive disease [PD], stable disease [SD], a partial response [PR] or a complete response [CR]) as validated by the Response Evaluation Criteria in Solid Tumors (RECIST) | Up to 2 years
  Ninety-five percent confidence interval for the response rate at the MTD will be constructed using the Wilson score method.

CONTACTS AND LOCATIONS:
Overall Officials: George Wilding, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States